CLINICAL TRIAL: NCT04883385
Title: Adherence Between Thromboprophylaxis Prescriptions and Guidelines During the Post-partum Period After the Institution of a Local Protocol
Brief Title: Thromboprophylaxis by Low Molecular Heparin During the Post-partum Period
Acronym: THROM-PP2021
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0016
Record Dates: First submitted 2021-05-05; First posted 2021-05-12 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Thromboembolic Disease
Keywords: Thromboembolic disease; Thromboprophylaxis; Post-partum period; Pregnancy; low molecular heparin
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: medical data collection — collection of medical data from patients' medical records

SUMMARY:
The purpose of this study is to determine the current level of adequacy of the thromboprophylaxis prescriptions with the specific institutional protocol during the post-partum period. The institutional protocol is based on national and international guidelines.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) became the 4th cause of maternal mortality and the 2nd direct cause of maternal mortality in France.

The re are only few randomized studies on the thromboprophylaxis during the post-partum period. This expose some discrepancy between French guidelines, French Society of Anesthesia & Intensive Care Medecine (SFAR) and National College of French Gynecologists and Obstetricians (CNGOF ).

The duration and adequate dose of low molecular heparin prescriptions are unclear.

The level of adequacy of thromboprophylaxis prescriptions at Centre Hospitalier Sud Francilien with the SFAR recommendations appears to be less than 50 % in a preliminary unpublished study.

Since this assessment, institutional protocol synthesizing thromboprophylaxis guidelines during the post-partum was exposed and validated among medical staff (both anaesthesiologists ang obstetricians).

ELIGIBILITY:
Inclusion Criteria:

* >18 ages
* Who had given birth at Centre Hospitalier Sud Francilien
* Hospitalized during the puerperium at Centre Hospitalier Sud Francilien
* Being informed of the clinical trial and had offered any opposition for data collection

Exclusion Criteria:

* Curative treatment of thrombosis by Low molecular-weight or unfractioned heparin during pregnancy or post-partum period
* Curative anticoagulant therapy for any cause

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All patients who had given birth at Centre Hospitalier Sud Francilien
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-07-09 (Actual)

PRIMARY OUTCOMES:
Level of adequacy of the thromboprophylaxis prescriptions with the specific institutional protocol during the post-partum period | at one year
  Level of adequacy of the thromboprophylaxis prescriptions with the specific institutional protocol during the post-partum period

SECONDARY OUTCOMES:
Level of adequacy of the thromboprophylaxis prescriptions with the specific institutional protocol after spontaneous or induced vaginal delivery. | at one year
  Level of adequacy of the thromboprophylaxis prescriptions with the specific institutional protocol after spontaneous or induced vaginal delivery.
Level of adequacy of the thromboprophylaxis prescriptions with the specific institutional protocol after a elective or urgent caesar section | at one year
  Level of adequacy of the thromboprophylaxis prescriptions with the specific institutional protocol after a elective or urgent caesar section
causes of non-compliant prescriptions with the institutional protocol. | at one year
  Identify the causes of non-compliant prescriptions with the institutional protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Elsa BROCAS, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No